CLINICAL TRIAL: NCT04729361
Title: CGH-array in Prenatal Diagnosis of Isolated Severe and Early Intra-uterine Growth Restriction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Matthieu DAP, medical doctor (MD), Central Hospital, Nancy, France
Other Study IDs: 2021PI007
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: IUGR; Prenatal Disorder; Genetic Disease
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: CGH array analysis — CGH array analysis

SUMMARY:
According to french recommandations for IUGR management we have to propose a CGH-array analysis if the IUGR is severe (bellow the 3rd percentile) and early (in the second trimester). However there is no data to support this point of view.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* fetus with an isolated intra-uterine growth restriction (IUGR) severe (bellow the third percentile on CFEF curves) and early (between 21 and 24 gestational weeks).

Exclusion Criteria:

* associated IUGR (with other abnormalities during prenatal screening)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: fetus with an isolated intra-uterine growth restriction (IUGR) severe (bellow the third percentile on CFEF curves) and early (between 21 and 24 gestational weeks).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-31 (Estimated); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
rate of abnormal CGH-array in the groupe "severe and early" UGR | one-time (at the time of the analysis)